## טופס הסכמה

## תכנית התערבות בתיווך הורים לקידום מיומנויות שפתיות ורגש חיובי משותף

המחקר הנוכחי עוסק בהתערבות בתיווך הורים לקידום מיומנויות שפה ורגש חיובי משותף בקרב ילדים על הספקטרום האוטיסטי או בסיכון גבוה לאבחון. הילדים יקבלו את ההתערבות קודם כל מהחוקרים, ולאחר מכן מההורים, אשר ילמדו מהחוקרים כיצד להעביר את שיטת ההתערבות.

במסגרת ההתערבות ההורים יקבלו הדרכה מובנית בקידום היכולות השפתיות והחברתיות של ילדם.

כחלק מההתערבות, הנכם מתבקשים למלא מספר שאלונים שיסייעו לנו לעקוב אחר התפתחותם של הילדים והתקדמותם בעקבות ההשתתפות בהתערבות.

בנוסף, המפגשים יהיו מצולמים לצורך המחקר, ומדריכ/ה שמנחה את צוות המחקר יצטרף לפגישות באמצעות פלטפורמת זום. לא יהיה שימוש בצילומים אלה, אלא לצורכי המחקר, גם לא לצרכי פרסום המחקר או כל סוג אחר של פרסום, <u>אלא אם הינך מסכימ/ה לכך במפורש בסעיף</u> המתאים לעיל.

כל המידע שייאסף בתהליך ישמר בסודיות תחת אבטחה מרבית וישומש רק לצרכי המחקר. ההשתתפות במחקר על בסיס התנדבותי, וזכותך להפסיק את השתתפותך בכל עת.

| יכימ/ה להשתתף בניסוי<br>לא | אני מס<br>כן |
|---|---|
| יי.<br>ישה לחוקרי המחקר להשתמש בצילומי הווידאו לצורכי פרסום והמחש<br>ר, ולצרכים אלו בלבד | אני מר |
| לא | כן |
| ת.ז | שם<br>חתימה |

לשאלות והבהרות ניתן לפנות לתמר מץ ויסמן, ביה"ס לחינוך ע"ש סימור פוקס:

tamar.matzvaisman@mail.huji.ac.il